CLINICAL TRIAL: NCT02629289
Title: A Phase 1 Study Assessing The Pharmacodynamic And Pharmacokinetic Equivalence Of HSP-130 With US-approved Neulasta (Registered) And EU-approved Neulasta (Registered) Administered As A Single Subcutaneous Dose To Healthy Volunteers
Brief Title: A Comparative Study to Evaluate the Effect of HSP-130, US-approved Neulasta and EU-approved Neulasta in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ZIN-130-1505; C1221001 (Other: Alias Study Number)
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2016-07-15 (Estimated); Status verified 2016-07

CONDITIONS: Neutropenia
Keywords: HSP-130; Pharmacodynamic and Pharmacokinetic equivalence; Pegfilgrastim
MeSH Terms: conditions — Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Other): HSP-130, 6 mg, single subcutaneous (SC) injection in the deltoid region
  Interventions: Drug: HSP-130
- Treatment B (Other): US-approved Neulasta, 6 mg, single SC injection in the deltoid region
  Interventions: Drug: US-approved Neulasta
- Treatment C (Other): EU-approved Neulasta, 6 mg, single SC injection in the deltoid region
  Interventions: Drug: EU-approved Neulasta

INTERVENTIONS:
Drug: HSP-130
  Other Names: Pegylated filgrastim
  Arms: Treatment A
Drug: US-approved Neulasta
  Other Names: Pegfilgrastim, Amgen
  Arms: Treatment B
Drug: EU-approved Neulasta
  Other Names: Pegfilgrastim, Amgen
  Arms: Treatment C

SUMMARY:
This study is for healthy participants. This study tests single dose of the research drug HSP-130 against two existing approved drugs United States - approved Neulasta and European Union-approved Neulasta.

DETAILED DESCRIPTION:
There will be 25 healthy participants in each of the six sequence groups. A total of 150 participants will be studied in one site in Australia. In addition to the 150 participants included, alternate subjects will be asked to come to the site on the day prior to when dosing is scheduled to begin. There will be 3 treatment options with 3 study dosing periods (1, 2 and 3) and at least 56 days between each treatment. The subject once asked to take part in the study will be assigned by chance (randomized) to one of the sequence groups as mentioned above (1, 2, 3, 4, 5, or 6).

ELIGIBILITY:
Inclusion Criteria:

1. Provides written informed consent approved by an Independent Ethics Committee (IEC) prior to any study related activities
2. Healthy male or female volunteers between 18 and 65 years of age (both inclusive)
3. Body mass index (BMI) between 19 and 30 kg/m^2, inclusive, and body weight of not <50 kg or >100 kg
4. Non-smoker (defined as a subject who has not smoked and has not used nicotine containing products for at least 3 months prior to study drug administration and has a negative urine screen for cotinine) at Screening
5. Female subjects of childbearing potential and male subjects and their partners of childbearing potential, agree to pregnancy prevention throughout the duration of the study (through the Follow-up Visit). Subjects and their partners must agree to use of an effective method of contraception, to avoid impregnation of females throughout the course of the study.

Subjects using oral contraceptives must be on a stable regimen for at least 3 months prior to Screening. Adequate forms of contraception to be used include hormonal contraceptives (oral, patch, depot), intrauterine devices (IUD), barrier contraceptive methods, such as diaphragm, cervical cap/shield, male condoms and female condoms.Sexually active subjects must use contraception while on study drug from admission to the Follow-up Visit. Male subjects must also refrain from donating sperm from admission to the Follow-up visit 6. Willing and able to comply with the requirements of the protocol and available for the planned duration of the study

Exclusion Criteria:

1. Any active systemic or immunologic disease or condition, including but not limited to the following general categories: cardiovascular/pulmonary, hepatorenal, or systemic infection, or lactation
2. History of, or current, malignancy with the exception of adequately treated squamous or basal cell carcinoma of the skin or cervical carcinoma in situ within 5 years
3. Any disease or condition that might interfere with the absorption, distribution, metabolism, or excretion of the study drug or would place the subject at increased risk
4. Hematologic laboratory abnormalities including leukocytosis (defined as total leukocytes >11,000/μL), leukopenia (defined as total leukocytes <4000/μL), neutropenia (defined as ANC <1500/μL) or thrombocytopenia (defined as platelet count of <150/μL)
5. Clinically significant, as judged by the investigator, vital sign or 12-lead ECG abnormality
6. History of biological growth factor exposure, including but not limited to filgrastim and other granulocyte-colony stimulating factors in the context of treatment, prophylaxis, peripheral blood stem cell mobilization, or previous investigational study setting. This also includes exclusion for history of interferon, epoetin, and intravenous immunoglobulin (IVIG) exposure
7. Receipt of live vaccination, or exposure to communicable viral diseases such as, varicella, mumps, or measles within the 4 weeks prior to Screening
8. Surgery within the 4 months prior to Screening
9. Use of any prescription medicine (with the exception of contraceptives) within 7 days or at least 5 half-lives, whichever is longer. Use of oral or parenteral anticoagulant or antiplatelet agents and corticosteroids should be specifically queried
10. Administration of a drug by depot injection (with exception of depot contraception) within 30 days prior to Randomization or 5 half-lives of that drug, whichever is longer
11. Use of over the counter medications, including aspirin and non-steroidal anti-inflammatory drugs, or natural preparations (dietary supplement or herbal product) within 7 days or at least 5 half-lives, whichever is longer. Vitamins and calcium are allowed (not to exceed 100% Daily Value)
12. History of drug or alcohol abuse within 2 years prior to Randomization, as determined by the investigator or a positive urine screen for drugs of abuse (UDS) at Screening. Screening for drugs of abuse will minimally include cannabinoids, opiates, barbiturates, amphetamines, cocaine, benzodiazepines, and alcohol
13. Drug sensitivity, allergic reaction to, or known hypersensitivity/idiosyncratic reaction to Escherichia coli-derived proteins, filgrastim, other granulocyte-colony stimulating factors, or pegylated agents
14. History of splenic rupture (or subject who is asplenic), pulmonary infiltrate or pneumonia, sickle cell disease, chronic neutropenia, thrombocytopenia, or vasculitis
15. Any clinically significant, as determined by the investigator, abnormal laboratory evaluations, including human immunodeficiency virus antibody (HIVAb), hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (HCVAb), and liver function including alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 1.5 the upper limit of normal taken at Screening. Negative HIVAb status will be confirmed at Screening and the results will be maintained confidentially by the study site
16. Donated or lost 475 mL or more blood volume (including plasmapheresis) or had a transfusion of any blood product within 3 months prior to Screening
17. Participated in another clinical research study with administration of investigational drug within 30 days prior to Randomization
18. Potentially not be able to comply with the requirements of this clinical trial, to communicate effectively with study personnel, or is considered by the Investigator, for any reason, to be an unsuitable candidate for the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Area under the effect versus time curve for absolute neutrophil count (ANC) from the time of dose administration to 288 hours after dose administration (AUECANC) | Within 1 hour prior to dose administration and at 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Maximum observed value for ANC (ANC_Cmax) | Within 1 hour prior to dose administration and at 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.

SECONDARY OUTCOMES:
Time of maximum value for ANC (ANC_Tmax) | Within 1 hour prior to dose administration and at 12, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Area under the serum pegylated filgrastim versus time curve from the time of dose administration to time infinity (AUC0-∞) | Within 1 hour prior to dose and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Maximum observed serum pegylated filgrastim concentration (Cmax) | Within 1 hour prior to dose and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Area under the serum pegylated filgrastim versus time curve from the time of dose administration to the time of last measurable concentration (AUC0-t) | Within 1 hour prior to dose and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Time to maximum serum pegylated filgrastim concentration (Tmax) | Within 1 hour prior to dose and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Elimination half-life (t1/2) | Within 1 hour prior to dose and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.
Elimination rate constant (λz) | Within 1 hour prior to dose and at 1, 2, 4, 6, 8, 10, 12, 16, 24, 48, 72, 96, 120, 144, 168, 192, 216, 240, 264, and 288 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- CMAX (a Division of IDT Australia Limited), Adelaide, South Australia, Australia

REFERENCES:
- [Derived] Moosavi S, Borema T, Ewesuedo R, Harris S, Levy J, May TB, Summers M, Thomas JS, Zhang J, Yao HM. PF-06881894, a Proposed Biosimilar to Pegfilgrastim, Versus US-Licensed and EU-Approved Pegfilgrastim Reference Products (Neulasta(R)): Pharmacodynamics, Pharmacokinetics, Immunogenicity, and Safety of Single or Multiple Subcutaneous Doses in Healthy Volunteers. Adv Ther. 2020 Jul;37(7):3370-3391. doi: 10.1007/s12325-020-01387-x. Epub 2020 Jun 10. PMID 32524499